CLINICAL TRIAL: NCT03399721
Title: A Clinical Investigation of Kinetic Oscillation Stimulation by the Chordate System S101 in the Treatment of Non Allergic Rhinitis
Brief Title: Investigation of Kinetic Oscillation Stimulation by the Chordate System S101 in the Treatment of Non Allergic Rhinitis
Acronym: KOSNAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chordate Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR008
Record Dates: First submitted 2018-01-09; First posted 2018-01-16 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2022-07

CONDITIONS: Nasal Congestion; Non-allergic Rhinitis
MeSH Terms: conditions — Nasal Obstruction; Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chordate S101 Active (Active Comparator): Active treatment With Device Chordate S101
  Interventions: Device: Chordate S101
- Chordate S101 Placebo (Placebo Comparator): Placebo treatment With Device Chordate S101
  Interventions: Device: Chordate S101 Placebo

INTERVENTIONS:
Device: Chordate S101 — Active treatment: The controller creates air-mediated kinetic oscillations with regulated pressure and frequency during a preset treatment time
  Arms: Chordate S101 Active
Device: Chordate S101 Placebo — Placebo treatment: Placebo treatment is similar to active treatment, but with no oscillations. It is difficult to discern any difference between active and placebo treatment.
  Arms: Chordate S101 Placebo

SUMMARY:
This is an interventional, multicenter, double-blind, placebo-controlled trial in which patients diagnosed with non-allergic rhinitis will be randomized to either intranasal stimulation, or placebo treatment with the Chordate System at two occasions.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, multi-center study in which patients diagnosed with non-allergic rhinitis will receive intranasal stimulation with the Chordate System at two occasions. Objectives are to evaluate the efficacy of the procedure in reducing disease specific symptoms such as nasal congestion, rhinorrhea, nasal itching and sneezing, but also to investigate the influence on quality of life, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with persistent (>12w) symptoms of non-allergic rhinitis dominated by nasal congestion (± secretion) for an average of at least 1 h per day for at least 5 days during a period of 14 days.
2. Having nasal congestion as major symptom, and a median nasal congestion score of at least 2 (scale 0-3)
3. Male or female 18 - 65 years
4. Judged by the Investigator as suitable for participation in the study without safety concerns based on medical history and physical examination.
5. Willing and able to provide written informed consent prior to participation in the clinical investigation
6. Willing and able to comply with all study related procedures

Exclusion Criteria:

1. Patients with Allergic rhinitis, demonstrated by either positive skin prick test, Phadiatop or RAST during the last year.
2. Ongoing respiratory tract infection including nasal cavity at inclusion
3. Systemic steroid treatment less than 4 weeks before the inclusion in the study
4. Patients with a history of nasal surgery like: septoplasty, cosmetic surgery, conchal surgery or any other nasal surgery except closed reposition for nasal fracture during last year
5. History of frequent nose bleeds or a condition that increases the risk of excessive bleeding
6. Pronounced anterior septal deviation or other significant nasal pathology at endoscopic examination
7. Current malignancy of any kind
8. Known allergy to polyvinylchloride or medicinal liquid paraffin
9. Any disease, condition (medical or surgical) or drug or alcohol abuse which, in the opinion of the investigator, might compromise the study results, or would place the patient at increased risk.
10. Any implant with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker, defibrillator, vagal neurostimulator, deep brain stimulation, spinal stimulator, bone growth stimulator, or cochlear implant or any other implant in the head-, and neck region.
11. Previous treated with radiation on the face, head or neck regions
12. Female patients who are pregnant or become pregnant at any time from inclusion of the study until end of the 8 week follow-up visit
13. Received study drug in a clinical trial for an investigational drug within the previous 30 days, or 5 half-lives, whichever is longer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Nasal congestion | 3 month
  The primary performance endpoint is the responder rate based on the change in the weekly median nasal congestion score (taken from Total Nasal Symptom Score (TNSS)) from baseline to the 3 month follow-up visit

CONTACTS AND LOCATIONS:
Locations (13):
- Czechia (3):
  - Charles University Faculty of Medicine in Hradec Králové, Hradec Králové
  - Hospital Pardubice, Pardubice
  - Charles University Motol University Hospital, Prague
- Finland (3):
  - Helsinki University Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere
- Aristotle University, Thessaloniki, Greece
- Italy (2):
  - Azienda Ospedaliera di Padova, Padua
  - Fondazione Policlinico A Gemelli, Rome
- Academisch Medisch Centrum Amsterdam, Amsterdam, Netherlands
- United Kingdom (3):
  - University Hospital Birmingham, Birmingham
  - James Paget University Hospital, Great Yarmouth
  - Guys Hospital, Greate Maze Pond, London